CLINICAL TRIAL: NCT00322127
Title: A Pilot Study of the Safety and Activity of Escalating Doses of AMD3100 to Mobilize CD34+ Cells in Healthy Volunteers
Brief Title: An Evaluation of Safety and Efficacy of Escalating Doses of AMD3100 to Mobilize CD34+ Cells in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 060156; 06-H-0156
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Healthy Volunteers
Keywords: Hematopoietic Stem Cells; Mobilization; CXCR4; SDF-1; Mozobil; Healthy Volunteer; HV
MeSH Terms: interventions — plerixafor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1 (Experimental): AMD3100 given as a single 240 g/kg dose followed 14-90 days later by a single 320 g/kg dose
  Interventions: Drug: AMD3100
- 2 (Experimental): AMD3100 given as a single 320 g/kg dose followed 14-90 days later by a single 400 g/kg dose
  Interventions: Drug: AMD3100
- 3 (Experimental): AMD3100 given as a single 400 g/kg dose followed 14-90 days later by a single 480 g/kg dose.
  Interventions: Drug: AMD3100
- 4 (Experimental): randomized to either receive 240 g/kg first followed by 480 g/kg after a washout period or 480 g/kg first followed by 240 g/kg after a washout period.
  Interventions: Drug: AMD3100

INTERVENTIONS:
Drug: AMD3100 — a 2 mL clear glass vial containing 1.7 mL of a sterile isotonic solution.

SUMMARY:
This study will determine how safely and well people can tolerate AMD3100 at larger than normal doses to mobilize CD34+ cells, (stem cells). AMD3100 is a new drug designed to mobilize stem cells for transplantation in cancer patients. It pushes those cells into the circulation, making it easier to collect them, and it temporarily increases the number of stem cells in a person's blood.

Patients ages 18 to 50 in good health and who are not pregnant or breastfeeding may be eligible for this study. They will undergo the following tests and procedures:

* History and physical examination
* Review of medications, including those prescribed and over-the-counter, as well as nutritional supplements
* Blood tests for liver, kidneys, and other functions; and for infections including hepatitis and AIDS
* Pregnancy test
* Electrocardiogram

On the day they receive AMD3100, patients will be admitted to the Clinical Center. They will receive two doses, injected under the skin, at intervals separated by 14 to 90 days. Dose levels are 240 and 320 micrograms/kg and 400 and 480 micrograms/kg. For 24 hours following the first AMD3100 administration, blood will be collected periodically through a plastic tube at amounts dependent on doses of AMD3100 given. If patients receive one of the two highest doses, their heart rhythm will be monitored continuously during the hospital stay. From 7 to 10 days following administration of AMD3100, patients will give blood samples to monitor the effects. The second dose of AMD3100 will be given 14 to 90 days after the first one. Patients will return to the Clinical Center for the same procedures as done previously, but the dose of the drug will be higher.

Risks involve side effects of AMD3100. In previous studies, patients who received the drug experienced a temporary increase in white blood cell counts. Serious side effects have included abnormally low platelet clot, abnormal heart rhythm, and low blood pressure. Patients will be carefully monitored for such effects.

DETAILED DESCRIPTION:
Peripheral blood progenitor cells (PBPC) have become the preferred source of hematopoietic stem cells for allogeneic transplantation because of technical ease of collection and shorter time required for engraftment. Traditionally, granulocyte-colony stimulating factor (G-CSF) has been used to procure the PBPC graft. Although regimens using G-CSF usually succeed in collecting adequate numbers of PBPC from healthy donors, 5%-10% of subjects will mobilize progenitor cells poorly and may require multiple large volume apheresis or bone marrow harvesting.

AMD3100 is a bicyclam compound that inhibits the binding of stromal cell derived factor-1 (SDF-1) to its cognate receptor CXCR4. CXCR4 is present on CD34+ hematopoietic progenitor cells and its interaction with SDF-1 plays a pivotal role in the homing of CD34+ cells in the bone marrow. Inhibition of the CXCR4-SDF-1 axis by AMD3100 releases CD34+ cells into the circulation, which can then be collected easily by apheresis. Recently, several reports have demonstrated that large numbers of progenitor CD34+ cells are rapidly mobilized in healthy volunteers following a single subcutaneous injection of AMD3100. The ability to collect a large quantity of PBPC's with a single injection of this drug makes this an attractive agent for mobilizing both autologous and allogeneic donors for hematopoietic stem cell transplantation.

A phase one dose escalating trial of AMD3100 in healthy donors done outside the NHLBI suggested the peak CD34+ mobilizing effects of this agent occurred at the 240 microgram/kg dose. Of note, no dose limiting toxicities were observed at the highest dose level of 320 mcg/kg. In two current trials at the NHLBI, AMD3100 has also proven to be well tolerated at the 240 mcg/kg dose, however, the progenitor CD34+ cell yield following a matched volume apheresis was lower compared to G-CSF mobilizations collected from the same healthy volunteers. More importantly, the number of CD34+ cells collected following one dose of AMD3100 has frequently been less than 3 x 10(6) CD34+ cells/kg, the previously defined minimal dose of progenitor cells required to optimize allogeneic hematopoietic stem cell transplantation outcomes. In addition, preliminary data from non-human primate studies suggest that higher doses of AMD3100 may improve CD34+ cell yield in an apheresis collection.

Based on these data, it is possible that inter-subject variability in CD34+ cell mobilization may have led investigators (in the prior phase I study) to prematurely terminate AMD3100 dose escalation based on the perception that CD34+ doses had peaked. We therefore propose this dose escalating study, designed to evaluate the safety and activity of AMD3100 when administered in escalating higher doses (240 microgram/kg dose, 320 microgram/kg dose 400 microgram/kg dose 480 microgram/kg dose). Activity will be evaluated by measuring the most effective dose of AMD3100 in mobilizing progenitor CD34 + cells into the circulation in healthy donors. To minimize inter-subject variability, we will administer two different doses of AMD3100 to each subject, evaluating the peak CD34+ cell count achieved after each dose. Separate cohorts of healthy volunteers will be evaluated for each dose escalation. The short half life and rapid wash-out of AMD3100 allows for this method of study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Ages greater than or equal to18 years and less than or equal to 50 years

Normal renal function: creatinine less than 1.5 mg/dl

Normal liver function: total bilirubin less than 1.5mg/dl, ALT and AST levels must be below the laboratory's high normal value.

Normal blood count:

WBC 3000-10000/mm(3)

Granulocytes greater than 1500/mm(3)

Platelets greater than 150,000/mm(3), and

Hemoglobin (females greater than 11.1 g/dl, males greater than 12.7 g/dl)

Antecubital veins must be adequate for peripheral access for phlebotomy (subject must be eligible for normal blood donation)

Ability to comprehend the investigational nature of the study and provide informed consent

EXCLUSION CRITERIA: ANY OF THE FOLLOWING:

Active infection or history of recurrent infection, hepatitis B and C (HBsAg, Anti-HCV), HIV and/or HTLV-1

History of autoimmune disease such as rheumatoid arthritis, systemic lupus erythematous

History of cancer within the past 5 years excluding basal cell or squamous cell carcinoma of the skin

History of any hematologic disorders including thromboembolic disease

History of cardiac disease such as uncontrolled hypertension, peripheral vascular disease, myocardial infarction, cardiac arrhythmias or related symptoms such as tachycardia, chest pain, shortness of breath which have required medical intervention or treatment or a Framingham coronary disease risk prediction score of greater than 10% 10 year CHD risk

History of cerebrovascular disease, transient ischemic attack, or stroke

Pregnant or lactating

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2006-06-14 (Actual); Primary Completion 2015-01-23 (Actual); Study Completion 2015-01-23 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability profile of AMD3100 when administered in escalating higher doses in humans. | all
  safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gyger M, Stuart RK, Perreault C. Immunobiology of allogeneic peripheral blood mononuclear cells mobilized with granulocyte-colony stimulating factor. Bone Marrow Transplant. 2000 Jul;26(1):1-16. doi: 10.1038/sj.bmt.1702464. PMID 10918400
- [Background] Srour EF, Leemhuis T, Brandt JE, vanBesien K, Hoffman R. Simultaneous use of rhodamine 123, phycoerythrin, Texas red, and allophycocyanin for the isolation of human hematopoietic progenitor cells. Cytometry. 1991;12(2):179-83. doi: 10.1002/cyto.990120213. PMID 2049974
- [Background] Bender JG, Unverzagt KL, Walker DE, Lee W, Van Epps DE, Smith DH, Stewart CC, To LB. Identification and comparison of CD34-positive cells and their subpopulations from normal peripheral blood and bone marrow using multicolor flow cytometry. Blood. 1991 Jun 15;77(12):2591-6. PMID 1710512
- [Derived] Pantin J, Purev E, Tian X, Cook L, Donohue-Jerussi T, Cho E, Reger R, Hsieh M, Khuu H, Calandra G, Geller NL, Childs RW. Effect of high-dose plerixafor on CD34+ cell mobilization in healthy stem cell donors: results of a randomized crossover trial. Haematologica. 2017 Mar;102(3):600-609. doi: 10.3324/haematol.2016.147132. Epub 2016 Oct 20. PMID 27846612
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-H-0156.html